CLINICAL TRIAL: NCT03317028
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of CS02 Tablet in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: CS02 vs Placebo With Metformin in Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS02-001; NCT03308695 (obsolete NCT alias)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: T2DM With Inadequate Glycemic Control

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- high dose of CS02 (Experimental): Subjects will receive 450mg of CS02 combined with a stable dose of metformin monotherapy.
  Interventions: Drug: CS02 tablet and placebo tablet
- middle dose of CS02 (Experimental): Subjects will receive 300mg of CS02 combined with a stable dose of metformin monotherapy.
  Interventions: Drug: CS02 tablet and placebo tablet
- low dose of CS02 (Experimental): Subjects will receive 150mg of CS02 combined with a stable dose of metformin monotherapy.
  Interventions: Drug: CS02 tablet and placebo tablet
- placebo control (Placebo Comparator): Subjects will receive placebo combined with a stable dose of metformin monotherapy.
  Interventions: Drug: CS02 tablet and placebo tablet

INTERVENTIONS:
Drug: CS02 tablet and placebo tablet — Subjects receive CS02 tablet or placebo tablet BID daily with a stable dose of metformin monotherapy of ≥ 1500 mg/day for 12 weeks treatment.

SUMMARY:
The objective of the study is to compare the efficacy and safety of 3 doses CS02 Tablet in combination with a stable dose of metformin monotherapy against CS02 PTM (placebo) Tablet in combination with a stable dose of metformin monotherapy over a 12 weeks treatment period in subjects with type 2 diabetes mellitus with inadequate glycemic control on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with diagnosis of type 2 diabetes mellitus at least 12 weeks prior to Visit 1;
2. Outpatient, either male or female, aged 20 years or older from Taiwan and aged 18 years or older from united States; all subjects are ≤75 years old;
3. Subjects with a stable diet and exercise program for ≧8 weeks prior to Visit 1;
4. Subjects with HbA1c value ≧7.0% and ≦10.0% at Visit 1;
5. Subjects with a stable dose of metformin monotherapy of ≥1500 mg/day at least 12 weeks before randomization (Visit 2);
6. Body mass index (BMI) between 20.0 and 45.0 kg/m2at Visit 1;
7. Subjects have adequate liver function, defined as serum total bilirubin≤1.5 times the upper limit of normal (uLN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤3 times uLN at Visit 1;
8. Subjects have estimated glomerular filtration rate (e-GFR)* values of≧ 45ml/min/1.73m2 at Visit1;
9. Female subjects of childbearing potential， defined as women≤ 55 years old or history of amenorrhea ≤ 12 months prior to the study entry or not surgically sterile, must have a negative pregnancy test at Visit 1 and agree to use a highly effective contraceptive method during the study period;
10. Willing to provide a written informed consent form;
11. Willingness and ability to comply with treatment plans, scheduled visits, required laboratory tests, and other study procedures;

Exclusion Criteria:

1. Subjects with type 1 diabetes mellitus, secondary diabetes mellitus, or gestational diabetes;
2. Subjects with acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma at Visit 1 or Visit 2;
3. Subjects with hypotension (average systolic pressure < 90 mm Hg*) at Visit 1 or Visit 2;
4. Subjects with cardiogenic shock within 8 weeks prior to Visit 1;
5. Subjects with sick sinus syndrome, second- or third-degree atrioventricular block (AV block);
6. Subjects with atrial flutter or atrial fibrillation and an accessory bypass tract (e.g., Wolff-Parkinson-White, Lown-Ganong-Levine syndromes);
7. Subjects with recurrence or history of transient ischemic attack or coronary artery bypass surgery;
8. Subjects with history of cerebrovascular attack, myocardial infarction, serious cardiac disease (New York Heart Association NYHA Class III to IV), left ventricular ejection fraction≦40% within 12 weeks prior to Visit 1, or those with cardiovascular disease or cerebrovascular disease that may affect the administration of IP tablets (CS02) or its safety assessment in the opinion of the investigator or sub-investigator;
9. Female subjects who are nursing or pregnant during the study period;
10. Subjects are on a weight loss program and not in the maintenance phase or have started a weight loss medication including but not limited to Orlistat, Phentermine, Osymia, or Belviq or have undergone bariatric surgery within 8 weeks prior to Visit 1 or any type of surgery planned during the study;
11. Subjects with a clinically severe gastrointestinal disorder including diabetic gastroparesis; irritable bowel disease; recurrent episodes of nausea, vomiting, diarrhea and abdominal pain within 12 weeks prior to Visit 1;
12. Subjects have a history or current of substance or alcohol abuse;
13. Subjects have uncontrolled psychiatric disorder(s);
14. Subjects are less than 5 years free of malignancy (except for cured basal cell carcinoma of skin and cured carcinoma in situ of the uterine cervix);
15. Subjects have participated in another clinical trial within the last 12 weeks prior to Visit 1;
16. Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments, or inappropriate for inclusion per investigators, judgments;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
The HbA1c treatment effect among CS02 groups and the Placebo group | 12 weeks
  To assess 208 evaluable subject of the change in HbA1c from baseline to end of treatment among CS02 groups and CS02 placebo to match group will be compared with the analysis of covariance model including baseline HbA1c as covariate, and treatment groups and regions as fixed effects.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Applied Research Center of Arkansas, Inc., Little Rock, Arkansas
  - Clinical Research of South Florida, Coral Gables, Florida
  - The Community Research of South Florida, Hialeah, Florida
- Taiwan (10):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans general Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital_Linkou, Taoyuan District

REFERENCES:
- [Derived] Wang CY, Huang KC, Lu CW, Chu CH, Huang CN, Chen HS, Lee IT, Chen JF, Chen CC, Chen CS, Hsieh CH, Tien KJ, Chien HY, Huang YY, Hsu JP, Shane GT, Chang AC, Wu YC, Sheu WH. A Randomized Controlled Trial of R-Form Verapamil Added to Ongoing Metformin Therapy in Patients with Type 2 Diabetes. J Clin Endocrinol Metab. 2022 Sep 28;107(10):e4063-e4071. doi: 10.1210/clinem/dgac436. PMID 35917580